CLINICAL TRIAL: NCT04115904
Title: Acute Pain Rate of Single Versus Two-visit Root Canal Treatment of Teeth With Necrotic Pulp and Apical Periodontitis: A Multicenter Clinical Trial
Brief Title: Acute Pain Rate of Single Versus Two-visit Root Canal Treatment of Teeth With Necrotic Pulps
Acronym: Acute pain
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universidad Autonoma de Baja California (Other)
Responsible Party: Principal Investigator, Jorge Paredes Vieyra, Dr. Jorge Paredes Vieyra DDS, MsC, PhD, Universidad Autonoma de Baja California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019
Record Dates: First submitted 2019-10-02; First posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Ibuprofen; Dental Implantation, Endosseous, Endodontic

STUDY DESIGN:
Intervention Model Description: 110 teeth with a diagnosis of pulp necrosis and apical radiolucency at the apex.Working length was established with EAL and confirmed radiographically. M4system with Flex-R files were used to complete canal preparation. Level ofdiscomfort were recorded and cases with severe postoperative pain
Who Masked: Investigator
Masking Description: compare Incidence of acute painafter single-visit ortwo-visits treatment of teeth with necrotic pulp
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post-endodontic Pain after a RCT (Experimental): Ibuprofen for Post operative pain. Take 400 mg takena week after. Incidence of flare ups after a single vsmultiple visits root canal treatments.
  Interventions: Procedure: Ibuprofen for post operative pain
- Acute pain (Experimental): Acetaminophen 325 mg for Acute pain. Taken secondday after. Incidence of Post operative pain after rootcanal treatment in one vs two visits
  Interventions: Procedure: Ibuprofen for post operative pain

INTERVENTIONS:
Procedure: Ibuprofen for post operative pain — All treatment sessions were approximately 45 minutes in length to allow for acceptable time for completionof treatment and retreatment in one or two visits. Allthe clinical procedures were performed by the author.Following local anesthesia with 2% lidocaine with1:100,000 epinephrine (Septodont Saint-Maur desFossés, France) and rubber dam isolation the toothwas disinfected with 5.25% NaOCl (Ultra bleach,Bentonville, AR, USA).
  Other Names: Endodontic therapy

SUMMARY:
Aim to compare acute pain rate after single-visit ortwo-visits treatment of teeth with necrotic pulp and apical periodontitis .90 teeth with a diagnosis of pulp necrosis and apical radiolucency at the apex.Working length was established with EAL and confirmed radiographically. Flex-R files were used to complete canal preparation. Level ofdiscomfort were recorded and cases with acute postoperative pain.

DETAILED DESCRIPTION:
90 teeth with a diagnosis of pulp necrosis and apical radiolucency at the apex.Working length was established with EAL and confirmed radiographically. M4system with Flex-R files were used to complete canal preparation. Level ofdiscomfort were recorded and cases with severe postoperative pain and/orswelling were classified as acute pain.

ELIGIBILITY:
Inclusion Criteria: a) Radiographic evidence of apical periodontitis (minimum size ≥2.0mm x 2.0 mm) and a diagnosis of pulpal necrosis confirmed by negativeresponse to hot and cold tests and b) Need for retreatment. Thermal pulptesting was performed by the author, and radiographic interpretation wasverified by one certified oral surgeon

-

Exclusion Criteria:

* patients without inclusion requirements or failure to obtain patient ́sauthorization. Patients, were excluded if they were younger than 18 yearsold, pregnant, had a positive history of antibiotic use within the past month,suffered from diabetes, or other systemic diseases. Teeth with periodontalpockets deeper than 4 mm also were excluded of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients from 18-65 years, both: male , fenale
Enrollment: 90 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2018-09-29 (Actual); Study Completion 2019-09-28 (Estimated)

PRIMARY OUTCOMES:
Pain intensity measure with general pain scale | a week
  Each patient will recall a week to evaluate post operative pain

CONTACTS AND LOCATIONS:
Locations (4):
- Mexico (4):
  - Jorge Paredes Vieyra, Tijuana, Baja Califronia
  - Jorge Paredes Vieyra, Tijuana, Estado de Baja California
  - Jose Clemente Orozco, Tijuana, Estado de Baja California
  - Jose Clemente, Tijuana, Estado de Baja California

IPD SHARING:
Plan to Share IPD: Yes
Each participant will be evaluated a week after the treatment
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Acute pain rate
Access Criteria: Evaluate the acute pain rate